CLINICAL TRIAL: NCT06974357
Title: Evaluation of Genetic Abnormalities Amongst Calcium Phosphate Predominant Stone Formers With Alkaline Urine pH on 24 Hour Urine Testing
Brief Title: Evaluation of Genetic Abnormalities Amongst Calcium Phosphate Stone Formers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ryan L Steinberg (Other)
Responsible Party: Sponsor-Investigator, Ryan L Steinberg, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 202503463
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Nephrolithiasis
Keywords: Urolithiasis; Calcium Phosphates; Genetics; Urine
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calcium Phosphate genetic testing (Experimental): drawing blood samples from patients in Urology clinic
  Interventions: Diagnostic Test: Genetic testing

INTERVENTIONS:
Diagnostic Test: Genetic testing — blood draws for genetic testing

SUMMARY:
Kidney stones continue to affect more and more people in the United States with the most recent estimate being 1 in 9 people will develop a stone in their life. While family history is a known risk factor for stone disease, it remains unclear whether this is related to learned dietary habits or a truly inheritable genetic condition. Known inheritable genetic conditions linked to stone formation are uncommon, and thus, routine genetic testing is not currently recommended by any major urologic organizations. Patients who form calcium phosphate predominant stones, a less common type of stone composition, tend to have alkaline urine pH which suggests that the kidneys are unable to rid the body of acid. Management of such patients for stone prevention can be difficult. The Iowa Institute for Human Genomics is one of only a handful of commercial labs which offers genetic testing for stone disease. The aim of this study is to assess the rate of genetic abnormalities amongst calcium phosphate predominant stone formers with alkaline urine. To this end, the investigators plan to enroll calcium phosphate predominant stone forming patients with alkaline urine on 24 hour urine collection who obtain their health care at UIHC to undergo free genetic testing via blood draw to assess for genetic abnormalities. The investigators will also collect information already available in the subject's chart to assess for other patterns between blood and urine tests and any genetic variants.

ELIGIBILITY:
Inclusion Criteria:

* Any patient, aged 18-90 and not incarcerated, under the care of a urologist at UIHC with known kidney stone composition including >=60% calcium phosphate and baseline 24 hour urine pH of >=6.3

Exclusion Criteria:

- Any patient over the age of 90 years old, incarcerated or without any evidence of calcium phosphate stone composition

* No struvite component on prior stone analysis
* No bacteria with urease producing organism at time of stone removal
* No history or evidence of systemic acidosis
* No use of acetazolamide, topiramate, zonisamide, valproic acid
* Stage >=3 CKD (GFR<60)
* Hepatic disease
* Pregnancy
* History of osteoporosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of genetic variants | 1 year
  assess the overall rate of genetic variants among the stone population

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No